CLINICAL TRIAL: NCT00520052
Title: Frequency of Zoledronic Acid to Prevent Further Bone Loss in Osteoporotic Patients Requiring Androgen Deprivation Therapy for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wirral University Teaching Hospital NHS Trust (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57/03
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Osteoporosis
Keywords: bisphosphonates, prostate cancer, bone density, osteoporosis
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LHRH Group (Active Comparator): Patients on LHRH agonists and zoledronic acid
  Interventions: Drug: zoledronic acid
- Bicalutamide Group (Active Comparator): Patients on Bicalutamide and zoledronic acid
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — 5 doses of 4mg iv given 3 monthly over one year (as infusion over 15 mins in 100 mls normal saline)
  Other Names: zometa

SUMMARY:
The aim of this study is to determine if 3 monthly infusions of zoledronic acid, given over one year, improves the bone mineral density in osteoporotic patients undergoing androgen deprivation therapy for prostate cancer

DETAILED DESCRIPTION:
Androgen Deprivation Therapy is the mainstay of treatment for advanced prostate cancer. However they are associated with accelerated bone loss, osteoporosis and fractures. Previous studied looking at the use of zoledronic acid have predominantly studied men with a normal or osteopenic bone mineral density. However, it has been shown that upto 40% of men presenting with prostate cancer have osteoporosis and it is these who are at most risk of osteoporotic fractures. Our aim was to evaluate the efficiency of zoledronic acid in 2 groups of osteoporotic patients, those undergoing treatment with LHRH agonists and with antiandrogens.Peripheral and axial bone densitometry will be used to measure percentage changes in bone mineral density over 3 years. The first year with the patients on LHRH or antiandrogen, the second year continuing with their androgen deprivation therapy and zoledronic acid. Then bone mineral density will be measured one year following the last infusion of zoledronic acid to ascertain the optimum frequency of administration.

The study will also involve monitoring serum and urine bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

* patients with locally advanced prostate cancer who progress from normal/ osteopenic bone mineral density to osteoporosis while on LHRH agonists (LHRH Group). Also patients who have been commenced on Bicalutamide due to osteoporosis at presentation (Bicalutamide Group)

Exclusion Criteria:

* patients with elevated prostate specific antigen, any illness or medication that would affect bone and mineral metabolism, previous bisphosphonate treatment, severe hepatic or renal insufficiency.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-08; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
axial and peripheral bone mineral density | over 3 years

SECONDARY OUTCOMES:
serum and urine bone turnover markers | over 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nigel J Parr, MBBS, FRCS, MD, Principal Investigator — Wirral Hospital University NHS Trust
Locations (1):
- Wirral Hospitals Universirt NHS Trust, Upton, Wirral, Merseyside, United Kingdom